CLINICAL TRIAL: NCT06165146
Title: A Phase I, Open-label, Fixed-sequence, Drug Interaction Study to Investigate the Effect of Multiple Oral Doses of Pirtobrutinib (LOXO-305) on the Pharmacokinetics of Repaglinide (CYP2C8 Substrate) in Healthy Subjects
Brief Title: A Study of the Effects of Pirtobrutinib (LOXO-305) on Repaglinide (CYP2C8 Substrate) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: LOXO-BTK-20016; J2N-OX-JZNL (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-11-30; First posted 2023-12-11 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — repaglinide; pirtobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Period 1: 0.5 mg Repaglinide (Experimental): Participants received a single oral dose of 0.5 milligrams (mg) repaglinide tablet, in the morning on Day 1.
  Interventions: Drug: Repaglinide
- Period 2: 200 mg Pirtobrutinib QD (Experimental): Participants received oral doses of 200 mg pirtobrutinib tablets, once daily (QD) in the morning from Day 2 to Day 11.
  Interventions: Drug: Pirtobrutinib
- Period 2: 200 mg Pirtobrutinib QD + 0.5 mg Repaglinide (Experimental): Participants received oral doses of 200 mg pirtobrutinib QD and 0.5 mg repaglinide tablets, in the morning on Day 12.
  Interventions: Drug: Repaglinide; Drug: Pirtobrutinib

INTERVENTIONS:
Drug: Repaglinide — Administered orally.
  Arms: Period 1: 0.5 mg Repaglinide; Period 2: 200 mg Pirtobrutinib QD + 0.5 mg Repaglinide
Drug: Pirtobrutinib — Administered orally.
  Other Names: LOXO-305; LY3527727
  Arms: Period 2: 200 mg Pirtobrutinib QD; Period 2: 200 mg Pirtobrutinib QD + 0.5 mg Repaglinide

SUMMARY:
The main purpose of this study is to evaluate the effect of pirtobrutinib (LOXO-305) on single oral dose of repaglinide (CYP2C8 substrate) when administered as multiple doses by conducting the blood tests to measure how much pirtobrutinib (LOXO-305) is in the bloodstream and how the body handles and eliminates pirtobrutinib (LOXO-305) in adult healthy participants. The study will also evaluate the safety and tolerability of pirtobrutinib (LOXO-305). The study is conducted in two periods. Participants will stay in this study for up to 54 days.

ELIGIBILITY:
Inclusion Criteria:

* Must have Body mass index (BMI) within the range of 18.0 to 32.0 kilograms per square meter (kg/m²), inclusive
* Male and female participants in good health, determined by no clinically significant findings from medical history, 12-lead Electrocardiogram (ECG), vital sign measurements, or clinical laboratory evaluations as assessed by the investigator
* Female participants of non-childbearing potential and male participants who follow standard contraceptive methods
* Must have comply with all study procedures, including the 16-night stay at the Clinical Research Unit (CRU) and follow-up phone call

Exclusion Criteria:

* History or presence of any diseases or conditions of clinical significance by the Investigator (or designee) and/or Sponsor
* Known ongoing alcohol and/or drug abuse within 2 years prior to Screening
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Unit, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 16 participants were enrolled in two period. In Period 1, participants received repaglinide only and in Period 2, participants received pirtobrutinib only followed by pirtobrutinib + repaglinide.
Period: Period 1 (Day 1)
Arm/Group | Period 1: 0.5 mg Repaglinide | Period 2: 200 mg Pirtobrutinib QD | Period 2: 200 mg Pirtobrutinib QD + 0.5 mg Repaglinide
Started | 16 | 0 | 0
Completed | 16 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Washout Period (11 Days)
Arm/Group | Period 1: 0.5 mg Repaglinide | Period 2: 200 mg Pirtobrutinib QD | Period 2: 200 mg Pirtobrutinib QD + 0.5 mg Repaglinide
Started | 16 (A washout period of 11 days was maintained between the dose of repaglinide on Day 1 and Day 12.) | 0 | 0
Completed | 16 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Period 2 (Day 2 to 11)
Arm/Group | Period 1: 0.5 mg Repaglinide | Period 2: 200 mg Pirtobrutinib QD | Period 2: 200 mg Pirtobrutinib QD + 0.5 mg Repaglinide
Started | 0 | 16 | 0
Completed | 0 | 16 | 0
Not Completed | 0 | 0 | 0
Period: Period 2 (Day 12)
Arm/Group | Period 1: 0.5 mg Repaglinide | Period 2: 200 mg Pirtobrutinib QD | Period 2: 200 mg Pirtobrutinib QD + 0.5 mg Repaglinide
Started | 0 | 0 | 16
Completed | 0 | 0 | 16
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Period 1: 0.5 mg Repaglinide: Participants received a single oral dose of 0.5 mg repaglinide tablet, in the morning on Day 1.
Arm/Group | Period 1: 0.5 mg Repaglinide
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (9.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration-time Curve, From Time 0 to the Last Measurable Concentration (AUC0-t) of Repaglinide
Description: PK: AUC(0-t) of repaglinide was reported.
Time Frame: Period 1, Day 1 (Pre-dose, 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10, 12, 16 and 24 hours post-dose); Period 2, Day 12 (Pre-dose, 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10, 12, 16 and 24 hours post-dose)
Population: The PK Population included all participants who received a dose of Repaglinide, had at least 1 quantifiable plasma concentration, and for whom at least 1 PK parameter was computed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Period 1: 0.5 mg Repaglinide | Period 2: 200 mg Pirtobrutinib QD + 0.5 mg Repaglinide
Number analyzed (Participants) | 16 | 16
hour*nanogram per milliliter (h*ng/mL) | 9.59 (36.9) | 22.2 (56.1)

2. Primary Outcome: PK: Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) of Repaglinide
Description: PK: AUC(0-inf) of repaglinide was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1: 0.5 mg Repaglinide | Period 2: 200 mg Pirtobrutinib QD + 0.5 mg Repaglinide
Number analyzed (Participants) | 16 | 16
h*ng/mL | 9.79 (36.5) | 22.5 (55.7)

3. Primary Outcome: PK: Percentage of AUC0-inf Extrapolated (AUC%Extrap) of Repaglinide
Description: PK: AUC-inf (%extrap) of repaglinide was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUC0-inf extrapolated
Arm/Group | Period 1: 0.5 mg Repaglinide | Period 2: 200 mg Pirtobrutinib QD + 0.5 mg Repaglinide
Number analyzed (Participants) | 16 | 16
percentage of AUC0-inf extrapolated | 1.94 (41.8) | 1.10 (60.6)

4. Primary Outcome: PK: Maximum Observed Concentration (Cmax) of Repaglinide
Description: PK: Cmax of repaglinide was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Period 1: 0.5 mg Repaglinide | Period 2: 200 mg Pirtobrutinib QD + 0.5 mg Repaglinide
Number analyzed (Participants) | 16 | 16
nanogram per milliliter (ng/mL) | 6.88 (59.3) | 13.6 (47.4)

5. Primary Outcome: PK: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Repaglinide
Description: PK: Tmax of repaglinide was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Period 1: 0.5 mg Repaglinide | Period 2: 200 mg Pirtobrutinib QD + 0.5 mg Repaglinide
Number analyzed (Participants) | 16 | 16
hour | 0.625 [0.333 to 1.00] | 0.750 [0.500 to 1.00]

6. Primary Outcome: PK: Apparent Terminal Elimination Rate Constant (Lambda Z) of Repaglinide
Description: PK: Lambda Z of repaglinide was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: one per hour (1/h)
Arm/Group | Period 1: 0.5 mg Repaglinide | Period 2: 200 mg Pirtobrutinib QD + 0.5 mg Repaglinide
Number analyzed (Participants) | 16 | 16
one per hour (1/h)
  Participant 1: number analyzed (Participants) | 1 | 1
  Participant 1 | 0.128 | 0.152
  Participant 2: number analyzed (Participants) | 1 | 1
  Participant 2 | 0.130 | 0.150
  Participant 3: number analyzed (Participants) | 1 | 1
  Participant 3 | 0.228 | 0.151
  Participant 4: number analyzed (Participants) | 1 | 1
  Participant 4 | 0.0847 | 0.157
  Participant 5: number analyzed (Participants) | 1 | 1
  Participant 5 | 0.0809 | 0.139
  Participant 6: number analyzed (Participants) | 1 | 1
  Participant 6 | 0.126 | 0.141
  Participant 7: number analyzed (Participants) | 1 | 1
  Participant 7 | 0.138 | 0.247
  Participant 8: number analyzed (Participants) | 1 | 1
  Participant 8 | 0.219 | 0.0995
  Participant 9: number analyzed (Participants) | 1 | 1
  Participant 9 | 0.183 | 0.208
  Participant 10: number analyzed (Participants) | 1 | 1
  Participant 10 | 0.197 | 0.218
  Participant 11: number analyzed (Participants) | 1 | 1
  Participant 11 | 0.147 | 0.118
  Participant 12: number analyzed (Participants) | 1 | 1
  Participant 12 | 0.139 | 0.174
  Participant 13: number analyzed (Participants) | 1 | 1
  Participant 13 | 0.181 | 0.148
  Participant 14: number analyzed (Participants) | 1 | 1
  Participant 14 | 0.105 | 0.170
  Participant 15: number analyzed (Participants) | 1 | 1
  Participant 15 | 0.221 | 0.220
  Participant 16: number analyzed (Participants) | 1 | 1
  Participant 16 | 0.0966 | 0.325

7. Primary Outcome: PK: Apparent Systemic Clearance (CL/F) of Repaglinide
Description: PK: CL/F of repaglinide was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/h)
Arm/Group | Period 1: 0.5 mg Repaglinide | Period 2: 200 mg Pirtobrutinib QD + 0.5 mg Repaglinide
Number analyzed (Participants) | 16 | 16
Liter per hour (L/h) | 51.1 (36.5) | 22.2 (55.7)

8. Primary Outcome: PK: Apparent Plasma Terminal Elimination Half-life (t½) of Repaglinide
Description: PK: t½ of repaglinide was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Period 1: 0.5 mg Repaglinide | Period 2: 200 mg Pirtobrutinib QD + 0.5 mg Repaglinide
Number analyzed (Participants) | 16 | 16
hour | 4.86 (34.6) | 4.11 (30.0)

9. Primary Outcome: PK: Apparent Volume of Distribution (Vz/F) of Repaglinide
Description: PK: Vz/F of repaglinide was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Period 1: 0.5 mg Repaglinide | Period 2: 200 mg Pirtobrutinib QD + 0.5 mg Repaglinide
Number analyzed (Participants) | 16 | 16
Liter | 358 (39.3) | 131 (66.0)

10. Primary Outcome: PK: Area Under the Concentration-time Curve, From Time 0 to the Last Measurable Concentration (AUC0-t) of Pirtobrutinib
Description: PK: AUC0-t of pirtobrutinib was reported.
Time Frame: Period 2, Day 12 (Pre-dose, 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10, 12, 16, 24, 42, 78 and 100 hours post-dose)
Population: The PK Population included all participants who received a dose of pirtobrutinib, had at least 1 quantifiable plasma concentration, and for whom at least 1 PK parameter was computed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 2: 200 mg Pirtobrutinib QD + 0.5 mg Repaglinide
Number analyzed (Participants) | 16
h*ng/mL | 184000 (22.1)

11. Primary Outcome: PK: Area Under the Concentration-time Curve During a Dosing Interval (AUCtau) of Pirtobrutinib
Description: PK: AUCtau of pirtobrutinib was reported.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 2: 200 mg Pirtobrutinib QD + 0.5 mg Repaglinide
Number analyzed (Participants) | 16
h*ng/mL | 105000 (18.0)

12. Primary Outcome: PK: Maximum Observed Concentration (Cmax) of Pirtobrutinib
Description: PK: Cmax of pirtobrutinib was reported.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 2: 200 mg Pirtobrutinib QD + 0.5 mg Repaglinide
Number analyzed (Participants) | 16
ng/mL | 7220 (15.0)

13. Primary Outcome: PK: Concentration Observed at the End of the Dosing Interval (Ctrough) of Pirtobrutinib
Description: PK: Ctrough of pirtobrutinib was reported.
Time Frame: Period 2: 24-hour post-dose on Day 12
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 2: 200 mg Pirtobrutinib QD + 0.5 mg Repaglinide
Number analyzed (Participants) | 16
ng/mL | 3050 (21.8)

14. Primary Outcome: PK: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Pirtobrutinib
Description: PK: Tmax of pirtobrutinib was reported.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Median (Full Range); unit: hour
Arm/Group | Period 2: 200 mg Pirtobrutinib QD + 0.5 mg Repaglinide
Number analyzed (Participants) | 16
hour | 1.00 [0.500 to 5.00]

15. Primary Outcome: PK: Apparent Systemic Clearance (CL/F) at Steady State of Pirtobrutinib
Description: PK: CL/F at steady state of pirtobrutinib was reported.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/h)
Arm/Group | Period 2: 200 mg Pirtobrutinib QD + 0.5 mg Repaglinide
Number analyzed (Participants) | 16
Liter per hour (L/h) | 1.91 (18.0)

ADVERSE EVENTS:
Time Frame: Baseline up to 23 days
Description: All participants who received at least 1 dose of study drug (repaglinide and/or pirtobrutinib).
Groups:
- Period 2: 200 mg Pirtobrutinib QD: Participants received oral doses of 200 mg pirtobrutinib tablets, QD in the morning from Day 2 to Day 11.
Arm/Group | Period 1: 0.5 mg Repaglinide | Period 2: 200 mg Pirtobrutinib QD | Period 2: 200 mg Pirtobrutinib QD + 0.5 mg Repaglinide
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 2/16 | 6/16 | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: 0.5 mg Repaglinide (N=16) | Period 2: 200 mg Pirtobrutinib QD (N=16) | Period 2: 200 mg Pirtobrutinib QD + 0.5 mg Repaglinide (N=16)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/46/NCT06165146/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/46/NCT06165146/SAP_001.pdf